CLINICAL TRIAL: NCT05541302
Title: A Retrospective Registry Study to Evaluate Extended NeuroStar® TMS Therapy for Adults With Major Depressive Disorder (MDD)
Brief Title: Retrospective TMS Therapy for Adults With MDD
Status: Completed | Type: Observational
Sponsor: Neuronetics (Other)
Collaborators: Southern California TMS Center (Unknown); Brown University (Other); TMS of South Tampa (Unknown); Sheppard Pratt Health System (Other); Nashville NeuroCare Therapy (Unknown); NAMSA (Other); Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: 44-50018-000
Record Dates: First submitted 2022-09-07; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- 1-20 TMS sessions: PHQ 9 ratings during this treatment period
  Interventions: Device: TMS
- 21 - 29 TMS sessions: PHQ 9 ratings during this treatment period
  Interventions: Device: TMS
- 30 TMS Sessions: PHQ 9 ratings during this treatment period
  Interventions: Device: TMS
- 31-36 TMS Sessions: PHQ 9 ratings during this treatment period
  Interventions: Device: TMS
- extended treatment 36 and beyond: PHQ 9 ratings during this treatment period
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Transcranial Magnetic Stimulation

SUMMARY:
Examine change in the magnitude of antidepressant effects as a function of number of TMS sessions and to determine whether extended treatment courses, beyond 30 and beyond 36 TMS sessions, result in improved efficacy.

DETAILED DESCRIPTION:
The efficacy of TMS in major depressive disorder (MDD) has markedly improved since the pivotal sham-controlled trials. While this enhanced efficacy has been attributed to use of longer treatment courses, the impact of number of treatment sessions on efficacy has not been adequately evaluated. The study device is the Neuronetics, Inc. NeuroStar® TMS Therapy System (K160703, K201158).The study is a retrospective analysis of real-world data from commercial centers. The data will be gathered from the Neuronetics database called TrakStar which collects records of each patient's treatment. The data will be used only as applicable to the objectives of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. At least 18 years of age.
3. Treatment with NeuroStar TMS Therapy.
4. Treatment date of November 01, 2008 or later.
5. Patient received at least one treatment with NeuroStar TMS Therapy according to standardized NeuroStar TMS Therapy treatment protocols.
6. Primary diagnosis of Major Depressive Disorder (MDD) with no comorbid diagnosis.
7. PHQ-9 scores available at baseline (pre-treatment).
8. Moderate or greater depression prior to the initial treatment course with NeuroStar TMS Therapy, defined as baseline score on the Physician Health Questionnaire-9 (PHQ- 9) ≥ 10.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises patients who were treated with Extended NeuroStar TMS Therapy for MDD on or after November 8, 2008, and whose treatment information was entered in the Neuronetics TrakStar registry at one of the qualifying participating study sites, and for whom the pre-specified required data elements are available in the TrakStar registry and who satisfy each of the study inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 6456 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Primary Objective | 1 to > 36 sessions for acute treatment sessions or > 6 weeks.
  The primary objective of this study are to evaluate the changes in the Patient Health Questionnaire-9 (PHQ-9) total score.
  and the rating of Clinical Global Impression - Severity (CGI-S) score following application of extended NeuroStar TMS Therapy compared to baseline.
Primary Objective | 1 to > 36 sessions for acute treatment sessions or > 6 weeks.
  The primary objective of this study are to evaluate the rating of Clinical Global Impression - Severity (CGI-S) score following application of extended NeuroStar TMS Therapy compared to baseline.

IPD SHARING:
Plan to Share IPD: No